CLINICAL TRIAL: NCT01609842
Title: Hybrid Effectiveness-Implementation Study to Improve Clopidogrel Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDP 12-179
Record Dates: First submitted 2012-03-09; First posted 2012-06-01 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Cardiovascular Disease; Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; adherence
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome | interventions — Pharmacists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phone reminders and pharmacist (Experimental): An alerted inpatient pharmacist or a designated study team member will bring the clopidogrel medication to the patient who has received a coronary stent. The patient will return home and receive IVR refill reminder calls.
  Interventions: Other: Multifaceted Intervention with pharmacist and IVR
- Usual Care (Other): The sites will have no interaction with the study personnel. The investigators will use database information to compare with the intervention sites
  Interventions: Other: Multifaceted Intervention with pharmacist and IVR

INTERVENTIONS:
Other: Multifaceted Intervention with pharmacist and IVR — An alerted inpatient pharmacists will bring the clopidogrel medication to the patient who has received a stent. The patient will return home and receive IVR messages about the importance of their medication as well as a refill reminder call.

SUMMARY:
Percutaneous coronary intervention (PCI) is a common invasive cardiovascular procedure performed in the VA with over 13,000 procedures in FY10. Clopidogrel is a critical adjuvant therapy following PCI with stent placement and is generally recommended for up to 1 year following the procedure. Despite the evidence supporting clopidogrel use, studies both outside and within the VA suggest that poor adherence to clopidogrel is common. However, prior interventions targeting non-adherence have not specifically focused on clopidogrel adherence among PCI patients.

There are many potential reasons for early clopidogrel discontinuation that involve patient and healthcare system factors. Patients reported the following reasons for discontinuing clopidogrel within 1 month after drug-eluting stent (DES) implantation: 1) misunderstanding the intended treatment duration; 2) conflicting recommendations about intended duration; 3) cost of the medication; and 4) patients' own decision to stop. In contrast, patients who continued to take clopidogrel reported the following as helpful: 1) communication such as letters from their physician; and 2) receiving specific instructions on clopidogrel use. These findings suggest that there are specific interventions that can be implemented to improve clopidogrel adherence.

Multi-modal interventions that incorporate frequent follow-up, especially with pharmacists and use interactive voice response (IVR) technology have improved medication adherence. IVR technology is a computer-based telephone system which initiates calls, receives calls, provides information, and collects data from users. IVR is currently a mainstay in the VA where patients frequently interact with these automated systems to get clinic appointments and/or refill prescriptions. IVR as part of multi-modal interventions have been well received by patients, increased adherence to medications (e.g., statins), and improved clinical outcomes (e.g., blood pressure, diabetes symptoms, health status). In addition, the investigators have successfully used IVR as part of a multi-modal, multi-site intervention including pharmacists to improve blood pressure levels among hypertensive patients. Accordingly, the investigators have designed the intervention to improve clopidogrel adherence that builds on the investigators' prior work and other successful adherence interventions from the literature.

The investigators propose a hybrid effectiveness-implementation study of a multi-faceted intervention to improve clopidogrel adherence at VA PCI centers. The investigators will use the VA's Cardiovascular Assessment Reporting and Tracking (CART-CL), a uniform cath lab procedure reporting tool at all VA cath labs. The intervention consists of 4 components: a) an alert from CART-CL will be sent to an inpatient pharmacist prior to discharge that a patient has received a stent; b) a pharmacist will bring clopidogrel to the patient's bedside prior to hospital discharge as well as educate the patient on the importance of and adherence to clopidogrel following PCI; c) interactive voice response (IVR) calls will be made to patients prior to the time of clopidogrel refill to remind patients and to facilitate refills during follow-up; and d) a Patient Aligned Care Team (PACT) member will contact patients who delay filling clopidogrel.

DETAILED DESCRIPTION:
I. Hypotheses and Specific Aims

The main objective is to conduct a type 1 hybrid effectiveness/implementation study to test the effectiveness of a successfully-piloted, evidence-based, multi-faceted intervention to improve patient adherence to clopidogrel following PCI. The proposed study will test the hypothesis that a successfully-piloted, evidence-based, multi-faceted intervention targeting Veterans following PCI procedure improves adherence to clopidogrel, reduces bleeding, myocardial infarction, stroke, and mortality among these patients, and is cost-effective. The proposed intervention will be based on the Chronic Care Model and will build on the investigators' pilot work as well as will leverage the VA's CART-CL, a uniform cath lab procedure reporting tool at all VA cath labs. The study will be evaluated using the REAIM framework consisting of the following components, reach, effectiveness, adoption, implementation and maintenance. The intervention will adapt elements of prior successful intervention, including patient education, collaboration between cath lab clinicians and impatient/outpatient pharmacy teams, and telemonitoring via interactive voice response (IVR) technology. This type I hybrid effectiveness/implementation study will be tested at 16 sites randomized to intervention with an average of 90 patients per site per 6 month period versus usual care.

Specific Aims:

1. To evaluate current practices at VA PCI facilities (n=20) to enhance adherence to clopidogrel, both at hospital discharge and during longitudinal follow-up.
2. To implement the multi-faceted intervention at 16 total sites through 4 roll-out phases (4 sites during each roll-out) in a randomized stepped wedge trial design.
3. To assess barriers and facilitators to intervention implementation during each roll-out phase through semi-structured interviews and incorporate lessons learned from each roll-out phase into subsequent roll-out phases.
4. To determine the effectiveness of a successfully-piloted, evidence-based, multi-faceted intervention versus usual care for improving clopidogrel filling at hospital discharge and adherence to clopidogrel (primary outcomes).
5. To determine the effectiveness of a successfully-piloted, evidence-based, multi-faceted intervention versus usual care for reducing the combined cardiovascular endpoints of bleeding, myocardial infarction, stroke, and mortality (secondary outcomes).
6. To assess the incremental cost-effectiveness of the successfully-piloted, evidence-based, multi-faceted intervention compared with usual care.

II. Background and Significance:

The investigators have successfully piloted the intervention to improve clopidogrel adherence following PCI. The investigators developed a software application integrated within CART-CL that assessed whether patients fill their clopidogrel prescription at hospital discharge. If clopidogrel was not filled, patients were contacted to identify barriers to medication filling. During follow-up, automated telephone calls were sent to patients to educate them about the importance of medication adherence and to remind them to refill clopidogrel prior to the refill due date. The software application successfully identified all 15 patients enrolled in the pilot who underwent PCI and whether they filled clopidogrel at hospital discharge at 2 VAMCs. In qualitative interviews about the automated calls, all patients indicated that the refill reminder messages were helpful. A majority of participants indicated that they felt the education/support from the messages or participation in the study was helpful or would be helpful to others. A few patients shared that the messages also supported refilling other medications and reminding them to ask clarifying questions about other medications. Following the successful pilot, the investigators' next step is to test the effectiveness of the intervention and study the implementation process across a range of VA facilities.

Building on the prior work and evidence from the literature, the investigators have developed the intervention informed by the Chronic Care Model (CCM) which is a framework that uses clinical information systems to facilitate evidence-based quality improvement. The investigators will leverage CART-CL, IVR technology, patient self-management, and team-based care to foster efficient, productive interactions between activated patients and proactive clinical teams to improve clopidogrel adherence. Further the components of the intervention directly address many of the reasons that patients have highlighted as leading to early clopidogrel discontinuation.

This study will refine the current state of knowledge on improving medication adherence in multiple ways. First, it combines multiple interventions that have been separately shown to be effective in improving medication adherence and addresses causes of clopidogrel non-adherence identified by patients. Second, the intervention focuses on a novel setting (i.e., patients discharged following PCI and transitioning to outpatient care) in contrast to prior adherence interventions that have focused only on patients with stable chronic diseases (e.g., hypertension). Prior work by the investigators' group and others suggest that the immediate post-ACS period, and more generally transitions from the inpatient to the outpatient setting, are particularly 'vulnerable periods' for medication adherence. Yet prior interventions have not specifically targeted this setting. Third, the targeted medication in this study has demonstrated short-term benefits and where non-adherence can have immediate adverse outcomes (e.g., stent thrombosis). Prior studies have focused on medications (e.g., hypertension medications) where non-adherence leads to problems longer term rather than the short term. Fourth, the study utilizes existing resources (i.e., cardiac data systems integrated with the VA electronic health record, VA pharmacists and patient-aligned care teams) to implement the intervention, improving the feasibility of broader implementation. Prior adherence interventions have generally required significant additional resources and the majority of quality improvement interventions are not continued following the end of the research project. This proposal will extend the current state of knowledge on medication adherence by demonstrating that a successful intervention will need multiple evidence-based components, and designed with plans for implementation in mind. Finally, this study is being conducted as a type I hybrid implementation study and therefore includes extensive study of the implementation process, which will yield both contributions to implementation science and facilitate wider dissemination if the intervention is found to be effective.

Furthermore, the study will make two important contributions to implementation science. First, the investigators will integrate a structured survey, the organizational readiness to change assessment (ORCA), for use in the formative and summative evaluations (described further in the evaluation plan). The ORCA has previously been psychometrically validated and found to predict implementation effectiveness. However, it has not been previously tested as a tool to support implementation. Findings from this study will help us understand if and how the ORCA can be used to support other implementation projects, and will contribute to users' materials for the survey. Second, the investigators are using an innovative study design, a randomized stepped wedge design, and building-in iterative formative evaluation to guide implementation of the intervention at sites in subsequent cohorts. As far as the investigators know, this kind of iterative rollout design with planned formative evaluation has not been used in an effectiveness/implementation hybrid study. If it works as planned, and provides useful formative evaluation findings from early cohorts, it may represent an important adaptation of the hybrid design.

In terms of VA patient care, if the intervention is successful, it will increase adherence to clopidogrel by helping patients take their anti-platelet medication routinely as prescribed, the quality of cardiovascular care for Veterans since adherence to clopidogrel has been associated with reductions in cardiovascular morbidity and mortality following PCI, and the efficiency of care by using telephone calls and telemonitoring for communication with patients rather than clinic visits. This study will leverage the automated pharmacy system and tele-monitoring technology for which the VA is a nationally recognized leader. Further, the study will address an important gap in knowledge (i.e., how to improve adherence to clopidogrel medications following PCI) and the findings can inform future interventions to improve adherence to other chronic cardiovascular medications. Finally, since the study is designed to be implemented using existing personnel/staff and current national platforms (i.e., CART-CL and PACT teamlets), it will be generalizable to other VA Medical Centers and Veterans.

ELIGIBILITY:
Inclusion Criteria:

At the PCI sites, the investigators will include

* all patients undergoing PCI with either a bare-metal (BMS) or drug-eluting stent (DES) and are prescribed clopidogrel regardless of the intended treatment duration
* other potential anti-platelet medications (thienopyridines) used following PCI to accommodate changes in practice (e.g., prasugrel or ticagrelor or ticlopidine).
* all patients undergoing PCI and receiving clopidogrel at the randomized sites, regardless of gender, ethnicity or race. Based on data from the national CART Program, the investigators anticipate ~23% minorities (African American 16.8%, Hispanic 4.4%, Asian/American Indian 1.4%) and 3.1 women will be included in the study.

Exclusion Criteria:

The investigators will exclude

* sites with low PCI volume,
* less than 20 PCI procedures performed during the last fiscal year (n=3),

Ages: 18 Years to 91 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14573 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P. Michael Ho, MD PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (15):
- United States (15):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS, Jackson, Mississippi
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - Salem VA Medical Center, Salem, VA, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beste LA, Glorioso TJ, Ho PM, Au DH, Kirsh SR, Todd-Stenberg J, Chang MF, Dominitz JA, Baron AE, Ross D. Telemedicine Specialty Support Promotes Hepatitis C Treatment by Primary Care Providers in the Department of Veterans Affairs. Am J Med. 2017 Apr;130(4):432-438.e3. doi: 10.1016/j.amjmed.2016.11.019. Epub 2016 Dec 18. PMID 27998682
- [Background] McCreight MS, Lambert-Kerzner A, O'Donnell CI, Grunwald GK, Hebert P, Gillette M, Jneid H, Parashar A, Grossman PM, Helfrich C, Mavromatis K, Saket G, Ho PM. Improving anti-platelet therapy adherence in the Veterans Health Administration: A randomized multi-site hybrid effectiveness-implementation study protocol. Contemp Clin Trials. 2019 Feb;77:104-110. doi: 10.1016/j.cct.2018.12.005. Epub 2018 Dec 19. PMID 30576842
- [Background] Doll JA, Tang F, Cresci S, Ho PM, Maddox TM, Spertus JA, Wang TY. Change in Angina Symptom Status After Acute Myocardial Infarction and Its Association With Readmission Risk: An Analysis of the Translational Research Investigating Underlying Disparities in Acute Myocardial Infarction Patients' Health Status (TRIUMPH) Registry. J Am Heart Assoc. 2016 Jun 13;5(6):e003205. doi: 10.1161/JAHA.116.003205. PMID 27412898
- [Derived] Ho PM, O'Donnell CI, McCreight M, Bavry AA, Bosworth HB, Girotra S, Grossman PM, Helfrich C, Latif F, Lu D, Matheny M, Mavromatis K, Ortiz J, Parashar A, Ratliff DM, Grunwald GK, Gillette M, Jneid H. Multifaceted Intervention to Improve P2Y12 Inhibitor Adherence After Percutaneous Coronary Intervention: A Stepped Wedge Trial. J Am Heart Assoc. 2022 Jul 5;11(13):e024342. doi: 10.1161/JAHA.121.024342. Epub 2022 Jun 29. PMID 35766258

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled January 2014-March 2017 at 15 VA cardiac catheterization laboratory sites in 4 waves according to the study design protocol
Pre-assignment Details: The participants reported in the Control Arm/Group were all unique patients; they were assigned as follows: pre-intervention control (n=6,081), post-intervention control (n=2,917), and concurrent intervention controls (n=4,869); there was no overlap between the control groups.
Groups:
- Intervention: Patients at intervention sites who received the intervention during the period of enrollment
- Control: Patients who did not received the intervention
Period: Pre-Intervention Control
Arm/Group | Intervention | Control
Started | 0 | 6081 (Intervention sites patients prior to enrollment period who did not receive the intervention)
Completed | 0 | 6081
Not Completed | 0 | 0
Period: Post-Intervention Control
Arm/Group | Intervention | Control
Started | 0 | 2917 (Intervention sites patients after enrollment period ended who did not receive the intervention.)
Completed | 0 | 2917
Not Completed | 0 | 0
Period: Concurrent Intervention Control
Arm/Group | Intervention | Control
Started | 708 | 4869 (Nonintervention sites patients during the period prior and post enrollment at the intervention sites)
Completed | 706 | 4869
Not Completed | 2 | 0
Not completed — pharmacy data not available | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-Intervention Control: Patients at intervention sites prior to the period of enrollment who did not received the intervention
- Post-Intervention Control: Patients from intervention sites after the period of enrollment ended and who did not receive the intervention
- Concurrent Intervention Control: Patients at nonintervention sites during the period of enrollment at the intervention sites
- Total: Total of all reporting groups
Arm/Group | Intervention | Pre-Intervention Control | Post-Intervention Control | Concurrent Intervention Control | Total
Number analyzed (Participants) | 706 | 6081 | 2917 | 4869 | 14573
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (9.1) | 66.4 (8.8) | 67.4 (8.9) | 66.4 (8.7) | 66.63 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 111 | 62 | 95 | 287
  Male | 687 | 5970 | 2855 | 4774 | 14286
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 82 | 28 | 32 | 146
  Asian | 2 | 21 | 4 | 13 | 40
  Native Hawaiian or Other Pacific Islander | 3 | 44 | 19 | 57 | 123
  Black or African American | 120 | 1028 | 597 | 584 | 2329
  White | 577 | 4906 | 2269 | 4183 | 11935
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Adherent Patients
Description: Percentage of patients whose clopidogrel prescription is filled at hospital discharge following the PCI stent placement as well as the percentage of patients who are adherent based on the pharmacy refill data in the year after hospital discharge. We used mixed logistic regression models for clopidogrel adherence (y/n PDC > 80%) as planned.
Time Frame: 12 months post PCI discharge
Measure: Count of Participants; unit: Participants
Groups:
- Concurrent Intervention Control: Patients at nonintervention sites during the period for patients prior to enrollment and post enrollment at the intervention sites
Arm/Group | Intervention | Pre-intervention Control | Post-intervention Control | Concurrent Intervention Control
Number analyzed (Participants) | 706 | 6081 | 2917 | 4869
Participants | 590 | 4484 | 2209 | 3633

2. Primary Outcome: Percentage of Participants With Anti-Platelet Medication Delay
Description: Percentage of Participants with Anti-Platelet Medication Delay. Delay is defined as filling anti-platelet medication >1 day after PCI discharge and not filling the anti-platelet medication prescription by the refill date
Time Frame: 12 months post PCI discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Pre-Intervention Control | Post-Intervention Control | Concurrent Intervention Control
Number analyzed (Participants) | 706 | 6081 | 2917 | 4869
Participants | 35 | 459 | 210 | 578

3. Primary Outcome: Mean PDC
Description: Proportion of days covered. The number of days that the patient had a pill to take divided by the number of days of follow-up (follow-up terminated at death or at 365 days).
Time Frame: 12 months post PCI discharge
Measure: Mean (Standard Deviation); unit: proportion of days covered
Arm/Group | Intervention | Pre-intervention Control | Post-intervention Control | Concurrent Intervention Control
Number analyzed (Participants) | 706 | 6081 | 2917 | 4869
proportion of days covered | 0.912 (0.172) | 0.851 (0.231) | 0.867 (0.217) | 0.858 (0.232)

4. Secondary Outcome: Hospitalizations
Description: Number of participants with hospitalizations
Time Frame: 12 months post PCI discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Pre-intervention Control | Post-intervention Control | Concurrent Intervention Control
Number analyzed (Participants) | 706 | 6081 | 2917 | 4869
Participants | 99 | 792 | 387 | 603

5. Secondary Outcome: Mortality
Description: Mortality
Time Frame: 12 months post PCI discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Pre-intervention Control | Post-intervention Control | Concurrent Intervention Control
Number analyzed (Participants) | 706 | 6081 | 2917 | 4869
Participants | 34 | 399 | 193 | 266

ADVERSE EVENTS:
Time Frame: 12 months post PCI discharge
Description: Only mortality data and serious adverse events collected; Other/Not Serious Adverse Events were not monitored/collected for the Intervention Arm/Group or Usual Care Arm/Group.
Groups:
- Intervention Arm: An alerted inpatient pharmacist or a designated study team member will bring the clopidogrel medication to the patient who has received a coronary stent. The patient will return home and receive IVR refill reminder calls.
  Multifaceted Intervention with pharmacist and IVR: An alerted inpatient pharmacists will bring the clopidogrel medication to the patient who has received a stent. The patient will return home and receive IVR messages about the importance of their medication as well as a refill reminder call.
Arm/Group | Intervention Arm | Usual Care
All-Cause Mortality (participants affected / at risk) | 34/706 | 858/13867
Serious Adverse Events (participants affected / at risk) | 99/706 | 1782/13867
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=706) | Usual Care (N=13867)
Reported hospitalizations of the participants (Cardiac disorders) | 3 (3) | 0 (0)
Reported hospitalizations of the participants (Gastrointestinal disorders) | 2 (2) | 0 (0)
Reported hospitalizations of the participants (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Reported hospitalizations of the participants (Renal and urinary disorders) | 6 (6) | 0 (0)
Reported hospitalizations of the participants (Infections and infestations) | 3 (3) | 0 (0)
Reported hospitalizations of the participants (General disorders) | 4 (4) | 0 (0)
Reported hospitalizations of the participants (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Other hospitalizations (General disorders) | 75 | 1782

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT01609842/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT01609842/SAP_000.pdf